CLINICAL TRIAL: NCT00876473
Title: The CPAP in Patients Affected by Acute Respiratory Failure
Brief Title: Evaluation of Different Continuous Positive Airway Pressure (CPAP) Systems in Patients With Acute Respiratory Failure
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: 590
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Acute Respiratory Failure
Keywords: CPAP; Acute Respiratory Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Acute Respiratory Failure patients
  Interventions: Procedure: CPAP system

INTERVENTIONS:
Procedure: CPAP system — Evaluating the effects of different CPAP systems on respiratory mechanics, respiratory effort and gas-exchange
  CPAP systems:
  Continuous high-flow CPAP with fixed value PEEP valve
  Continuous high-flow CPAP with Boussignac valve
  Demand flow CPAP supplied by ventilator

SUMMARY:
The aim of this study is to evaluate the performance, the tolerability and the efficacy on gas-exchange of different CPAP (Continuous Positive Airway Pressure) systems.

DETAILED DESCRIPTION:
Three CPAP systems are studied for each patient at the same level of PEEP: 1) continuous high-flow CPAP with fixed value PEEP valve; 2) continuous high-flow CPAP with Boussignac PEEP valve; 3) demand flow CPAP, supplied by a ventilator.

ELIGIBILITY:
Inclusion Criteria:

* Intubated-tracheostomized subjects receiving CPAP during the weaning from invasive mechanical ventilation

Exclusion Criteria:

* Hemodynamic instability
* Barotrauma
* Severe myopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Critically ill patients affected by Acute Respiratory Failure
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Respiratory mechanics, work of breathing, end-expiratory lung volume (EELV) and gas exchange | 30 minutes

SECONDARY OUTCOMES:
Comfort of breathing | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy